CLINICAL TRIAL: NCT06842277
Title: Reconstruction of Deficient Interdental Papilla Using Albumin-platelets Rich Fibrin- A Case Series
Brief Title: Treatment of Deficient Interdental Papilla Using Albumin-platelets Rich Fibrin
Acronym: A case series
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Salah Eldin Mahmoud Radwan, Master Student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20124
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Interdental Papilla Reconstruction; Deficient Interdental Papilla
Keywords: Reconstruction of deficient interdental papilla using injectable albumin platelets rich fibrin

STUDY DESIGN:
Intervention Model Description: A case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients whose had deficient interdental papilla (Other): treatment of patients whose had deficient interdental papilla using injectable Albumin -platelets rich fibrin
  Interventions: Biological: Injectable albumin platelets rich fibrin

INTERVENTIONS:
Biological: Injectable albumin platelets rich fibrin — Using injectable albumin platelets rich fibrin which is minimally invasive non surgical technique with autogenous , slow degradable and rich in leukocytes and growth factors material .

SUMMARY:
The goal of this ( A case series, clinical trial ) is treatment of deficient interdental papilla in patients who have interdental papillary loss class 1 or 2 in maxillary or mandibular anterior region with plaque index and gingival index less than 1 and the selected sites had distance between contact point and inter proximal bone crest less than 7mm and probing depth less than 4mm.

Hypothesis:

Albumin-PRF is an efficient treatment of deficient interdental papilla. The primary outcome ( distance between the contact point and papillary tip will be measured by periodontal probe) The participants will practice good oral hygiene measures

DETAILED DESCRIPTION:
The goal of this ( A case series , clinical trial ) treating patients whose complaint from poor esthetics and unappealing black triangles inn anterior sextant using an autogenous , biocompatible material ( Albumin platelets rich fibrin).

The selected patients had well -aligned maxillary teeth, no caries, no proximal restoration, fixed prosthesis, or any orthodontic appliance, at least one class 1or 2 interdental papilla loss in maxillary or mandibular anterior regions and at selected sites, distance between contact point and inter proximal bone crest less than 7mm and probing depth less than 4mm.

Also patients had plaque index and gingival index less than 1. Patients whose had advanced periodontal problems (advanced bone and soft tissue loss), a systemic condition affect blood components and healing, smokers and Patients who are pregnant will be excluded.

For all patients, full mouth scaling and root planing will be done, measuring probing depth, taking periapical radiograph for the target sites and taking rubber base impression will be done.

Operation phase:

Then preparation of injectable Alb-PRF, 10ml of intravenous blood will be withdrawn from antecubital region and will be centrifuged using plastic tubes at 700g for 8 minutes. The denaturated albumin will be obtained by tempering the platelet poor plasma layer for 10 minutes at 75 degrees Celsius then the residual cells and the growth factors detected in the buffy coat (liquid PRF) will be mixed again with the cooled albumin gel to form injectable albumin PRF. Obtained injectable Alb-PRF will be filled in the insulin syringes to use in the selected sites immediately after anesthesia. The needle of the insulin syringe will be inserted 2-3 mm apical to the papilla tip directed coronally making an angle of 45 degree to the long axis of the tooth with its bevel facing apically.

Post-injection, papilla will be gently massaged in an incisal direction, for a minute using a gauze.

Post-operative phase:

Patients will be instructed to use a soft toothbrush coronal to the gingival margin and prevent the use of interdental aids at the treated region.

Patients will be kept under follow up at 3 and 6 months wherein clinical and photographic parameters will be recorded.

Primary outcome:

Distance between contact point and papilla tip (Height of black triangle)

Secondary outcomes:

Surface area of black triangle Patient Satisfaction Interproximal papillary levels

ELIGIBILITY:
Inclusion Criteria:

* Patients' complaint from poor esthetics and unappealing black triangles in anterior sextant.
* Patients had well -aligned maxillary teeth, no caries, no proximal restoration, fixed prosthesis, or any orthodontic appliance.
* Patients had at least one class 1or 2 interdental papilla loss in maxillary or mandibular anterior regions.
* Patients had at selected sites, distance between contact point and inter proximal bone crest less than 7mm and probing depth less than 4mm.
* Patients had plaque index and gingival index less than 1.

Exclusion Criteria:

* Patient had advanced periodontal problems (advanced bone and soft tissue loss).
* Patients had a systemic condition affect blood components and healing.
* Smoker patients.
* Patients who are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Distance between contact point and papilla tip (Height of black triangle) | 6 months
  The distances between the contact point and papilla tip will be measured clinically by a periodontal probe

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry , Cairo University, Giza, Giza Governorate
  - Faculty of Dentistry Cairo University, Giza, Giza Governorate